CLINICAL TRIAL: NCT05098522
Title: A Phase 2a, Randomized, Double-Blind, Placebo-Controlled, Parallel-Design, Allergen Challenge Trial of 6 Repeat Doses of IRL201104 in Adult Participants With Seasonal Allergic Rhinitis.
Brief Title: Allergen Challenge Trial of IRL201104 in Seasonal Allergic Rhinitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Revolo Biotherapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RVLO 121-05
Record Dates: First submitted 2021-09-30; First posted 2021-10-28 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-05

CONDITIONS: Seasonal Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal | interventions — IRL201104

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: IRL201104 (Experimental): IRL201104 IV on Day 1, Day 14, Day 28, Day 42, Day 56, Day 70
  Interventions: Drug: IRL201104
- Arm 2: Placebo (Placebo Comparator): Placebo IV on Day 1, Day 14, Day 28, Day 42, Day 56, Day 70
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: IRL201104 — lyophilised powder for reconstitution for IV dosing
  Arms: Arm 1: IRL201104
Drug: Placebo — Matching placebo for IRL201104
  Arms: Arm 2: Placebo

SUMMARY:
The purpose of this allergen challenge study is to assess the efficacy of IRL201104 compared with placebo in adult participants with seasonal allergic rhinitis.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18 to 65 years old, inclusive, at time of signing the informed consent form (ICF).
2. Body mass index within the range 19 to 30 kg/m2.
3. A clinical history of grass pollen-induced allergic rhinitis for at least 2 years with peak symptoms in May, June, or July.
4. A clinical history of moderate to severe rhinitis symptoms interfering with usual daily activities or with sleep as defined according to the ARIA classification of rhinitis (Bousquet, Khaltaev et al 2008)
5. A clinical history of rhinitis for at least 2 years requiring treatment with either antihistamines or nasal corticosteroids during the grass pollen season.
6. Positive skin prick test response, defined as wheal diameter greater than or equal to 5 mm, to Phleum pratense.
7. Positive specific IgE, defined as greater than or equal to IgE class 2 (0.7 kU/L), against Phleum pratense.
8. A positive response to the nasal allergen challenge with Phleum pratense, defined as an increase in TNSS greater than or equal to 5 points.
9. Agree to follow the contraception requirements of the trial as described in Appendix 7.

   Female participants must agree to use highly effective contraception as described in Appendix 7, or must be of non-childbearing potential. A woman is considered to be of non-childbearing potential if she meets one of the following criteria:
   1. post-menopausal (amenorrhea for at least 12 months, and follicle-stimulating hormone [FSH] tests at screening confirms post-menopausal status)
   2. has no uterus, ovaries or fallopian tubes. c. documentation of non-childbearing potential from a reproductive specialist.
10. The ability to give informed consent and comply with study procedures.
11. Venous access as appropriate for IV dosing, as judged by the investigator or delegate.

Exclusion Criteria:

1. A prebronchodilator forced expiry volume in 1 second (FEV1) less than 70% of the predicted value at the screening baseline visit.
2. Clinical history of persistent asthma requiring regular inhaled corticosteroids for > 4 weeks per year outside of the grass pollen season.
3. Clinical history of moderate - severe allergic rhinitis, according to the ARIA classification, caused by a perennial allergen to which the participant is regularly exposed.
4. Clinical history of moderate-severe allergic rhinitis, according to the ARIA classification, caused by tree pollen (those with mild intermittent symptoms not requiring regular treatment may be included).
5. History of emergency visit or hospital admission for asthma in the previous 12 months.
6. History of chronic obstructive pulmonary disease.
7. History of significant recurrent acute sinusitis, defined as 2 episodes per year for the last 2 years, all of which required antibiotic treatment.
8. History of chronic sinusitis, defined as sinus symptoms lasting greater than 12 weeks that includes 2 or more major factors or 1 major factor and 2 minor factors. Major factors are defined as facial pain or pressure, nasal obstruction or blockage, nasal discharge or purulence or discolored postnasal discharge, purulence in nasal cavity, or impaired or loss of smell. Minor factors are defined as headache, fever, halitosis, fatigue, dental pain, cough, ear pain, pressure, or fullness.
9. History of systemic disease affecting the immune system such as autoimmune diseases, immune complex disease, or immunodeficiency.
10. At randomization, current symptoms of, or treatment for, upper respiratory tract infection, acute sinusitis, acute otitis media, or other relevant infectious process; serous otitis media is not an exclusion criterion. Participants may be re-evaluated for eligibility after symptoms resolve.
11. Active malignancy at randomization.
12. Any tobacco smoking within the last 6 months or a history of greater than or equal to 10 pack years.
13. Previous treatment by immunotherapy with grass pollen allergen within the previous 5 years.
14. History of bleeding disorders or treatment with anticoagulation therapy.
15. History of anti-IgE monoclonal antibody treatment.
16. Ongoing systemic immunosuppressive treatment.
17. History of intolerance to the study therapy, rescue medications, or their excipients.
18. Pregnant or lactating women. For women of childbearing potential, a positive serum or urine pregnancy test.
19. The use of any investigational drug within 30 days of the screening visit.
20. The presence of any medical condition that the investigator deems incompatible with participation in the study.
21. Moderate or severe renal impairment (eGFR <60 mL/min/1.73 m2) or end stage renal disease.

23. Known or suspected immunosuppression, including history of invasive opportunistic infections (eg, history of or active tuberculosis, non-tuberculous mycobacterial infections, histoplasmosis, listeriosis, coccidioidomycosis, pneumocystosis, aspergillosis) despite infection resolution, or otherwise recurrent infections of abnormal frequency, or prolonged infections suggesting an immunocompromised status, as judged by the investigator. 24. Clinically relevant abnormal history, physical findings, ECG, or laboratory values at the pre-study screening assessment that could interfere with the objectives of the study or the safety of the volunteer. 25. Clinical contraindication to intradermal challenge (IDC), skin prick test (SPT), skin prick titration (SPT), or nasal allergen challenge (NAC), to include:

1. Previous anaphylactic reaction to grass pollen or extract excipients
2. Acute inflammation of the nose or paranasal sinuses
3. Severe and uncontrolled bronchial asthma or chronic obstructive pulmonary disease
4. Systemic immunotherapy
5. A generalised dermatological condition rendering it impracticable to perform SPT or IDC on unaffected skin.
6. Severe dermatographism
7. Unable to cease antihistamines/other interfering drugs (i.e. antidepressants)
8. Concomitant use of beta-blockers

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2021-11-04 (Actual); Primary Completion 2023-03-27 (Actual); Study Completion 2023-03-27 (Actual)

PRIMARY OUTCOMES:
The mean diameter of the Intradermal Challenge (IDC) Late Phase Response (LPR) on Day 84 measured 8 hours post-challenge after 10 weeks of treatment with IRL201104 compared with placebo. | Day 84
  An analysis of covariance (ANCOVA) will be performed

SECONDARY OUTCOMES:
The largest diameter (mm) of the IDC Early Phase Response (EPR) at 30 minutes after 10 weeks of treatment with IRL201104 compared with placebo | Day 84
  An analysis of covariance (ANCOVA) will be performed
Skin prick test EPR endpoint titration of Grass Soluprick after 10 weeks of treatment with IRL201104 compared with placebo. | Day 84
  An analysis of covariance (ANCOVA) will be performed
The weighted average of the TNSS per hour following NAC after challenge on Day 1 and day 84 of treatment with IRL201104 compared with placebo. | Day 84
  An analysis of covariance (ANCOVA) will be performed
Percent change in peak nasal inspiratory flow (PNIF) after the NAC on day 1 and day 84 of treatment with IRL201104 compared with placebo. | Day 84
  An analysis of covariance (ANCOVA) will be performed
Concentration of IRL20114 levels. | Day 56
  IRL201104 plasma levels will be summarized for each blood sample draw timepoint
Vital Signs: Blood pressure | Day 84
  Summary statistics, by and across randomized treatment group
Vital Signs: Pulse rate | Day 84
  Summary statistics, by and across randomized treatment group
Vital Signs: oral body temperature | Day 84
  Summary statistics, by and across randomized treatment group
Vital Signs: respiration rate | Day 84
  Summary statistics, by and across randomized treatment group
Treatment Emergent Adverse Events | Day 84
  Summary statistics, by and across randomized treatment group
Incidence of treatment-emergent antidrug antibody (ADA) responses | Day 84
  Tabulated and presented as the number and percentage of participants exhibiting the response within each treatment group
Safety Laboratory: Biochemistry | Day 84
  Glucose, liver function tests, urea, and electrolytes will be analysed by summary statistics, by and across randomized treatment group with data from Day 1, 56 and 84.
Safety Laboratory: Haematology | Day 84
  Full blood count variables will be analysed by summary statistics, by and across randomized treatment group with data from Day 1, 56 and 84.

CONTACTS AND LOCATIONS:
Overall Officials: Anoshie Ratnayake, MD, Study Director — Revolo Biotherapeutics
Locations (2):
- United Kingdom (2):
  - Hammersmith Medicines Research, London
  - King's College London, London